CLINICAL TRIAL: NCT05917483
Title: Evaluation of Mechanical Characteristics and Prevention From Overuse Injury of Tendons of Elite Athletes Using Dynamic Sonography
Brief Title: Evaluation of Mechanical Characteristics of Tendons of Athletes Using Sonography
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NTUH-REC 201812022RINC
Record Dates: First submitted 2023-06-04; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2019-01

CONDITIONS: Overuse Injury; Rotator Cuff Injuries
MeSH Terms: conditions — Cumulative Trauma Disorders; Rotator Cuff Injuries | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasonography — Collect shoulder rotator cuff tendon ultrasound image during isotonic motion

SUMMARY:
The investigators analyzed the strain of the rotator cuff tendon of baseball pitchers obtained using ultrasonography and compared the change in peak tendon strain before and after the regular season.

ELIGIBILITY:
Inclusion Criteria:

* Baseball pitchers in city baseball team

Exclusion Criteria:

* History of shoulder disorder or surgery

Ages: 21 Years to 33 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Baseball pitcher from city baseball team and actively participating season games
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Peak tendon strain | Two months
  The peak value of tendon strain during the isotonic motion estimated from ultrasound image sequence

CONTACTS AND LOCATIONS:
Locations (1):
- Tianmu Sports Park/ Baseball Stadium, Taipei, Taiwan